CLINICAL TRIAL: NCT00747344
Title: A Phase 3, Multicenter, Randomized, Double-blind, Placebo-controlled Study Evaluating the Efficacy and Safety of Ustekinumab in the Treatment of Korean and Taiwanese Subjects With Moderate to Severe Plaque-type Psoriasis
Brief Title: A Phase 3 Trial to Look at the Safety and Effectiveness of Ustekinumab in Korean and Taiwanese Subjects With Moderate to Severe Plaque-type Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centocor, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR015313
Record Dates: First submitted 2008-09-04; First posted 2008-09-05 (Estimated); Results first posted 2012-10-05 (Estimated); Last update posted 2013-03-29 (Estimated); Status verified 2013-03

CONDITIONS: Psoriasis
Keywords: Psoriasis; Psoriatic Arthritis; Ustekinumab; CNTO 1275
MeSH Terms: conditions — Psoriasis; Arthritis, Psoriatic | interventions — Ustekinumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo - Controlled Period (CP) (Placebo Comparator)
  Interventions: Drug: Placebo - Controlled Period (CP)
- Ustekinumab 45 mg - CP (Experimental)
  Interventions: Drug: Ustekinumab 45 mg - CP
- Placebo to ustekinumab 45 mg - after CP (Experimental)
  Interventions: Drug: Placebo to ustekinumab 45 mg - after CP
- Ustekinumab 45 mg - after CP (Experimental)
  Interventions: Drug: Ustekinumab 45 mg - after CP

INTERVENTIONS:
Drug: Placebo - Controlled Period (CP) — Placebo, Weeks 0-12
  Arms: Placebo - Controlled Period (CP)
Drug: Ustekinumab 45 mg - CP — Ustekinumab 45 mg, Weeks 0-12
  Arms: Ustekinumab 45 mg - CP
Drug: Placebo to ustekinumab 45 mg - after CP — Placebo at Weeks 0 and 4, then ustekinumab 45 mg at Week 12 and Week 16
  Arms: Placebo to ustekinumab 45 mg - after CP
Drug: Ustekinumab 45 mg - after CP — Ustekinumab 45 mg at Weeks 0 and 4, then placebo at Week 12 and ustekinumab 45 mg at Week 16
  Arms: Ustekinumab 45 mg - after CP

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Ustekinumab in the treatment of patients with moderate to severe psoriasis in South Korea and Taiwan.

DETAILED DESCRIPTION:
This is phase 3, multicenter, randomized, placebo-controlled double-blind, parallel study of subcutaneous injection of placebo and ustekinumab 45mg in Taiwanese and Korean patients with moderate to severe plaque psoriasis. Ustekinumab is an experimental medicine that is being tested to see if it may be useful in treating moderate to severe psoriasis. The patients will receive either ustekinumab or placebo at week 0 or week 4, and will be followed up through week 36. Patients who randomized (study drug assigned by chance) to placebo will cross over to ustekinumab 45mg group at week 12 and week 16 .The effectiveness of ustekinumab will be compared with placebo treated patients at week 12. Safety information will be collected through week 36. Patients randomized to ustekinumab will receive placebo at week 12 to maintain the blind and additional dose of 45mg at week 16. This study will be conducted in approximately 13 sites in South Korea and Taiwan and will include approximately 120 patients with approximately 60 patients in each country. This study is "blinded." This means that neither you nor your study doctor will know in which group you are placed. However, in case of medical emergency, your study doctor can quickly find out which treatment group you are in. You may get either ustekinumab or placebo (which looks like the medicine being studied but has no active ingredients) at the start of the study. All patients in the study will eventually receive Ustekinumab after week 12. Patients assigned to the ustekinumab will receive 45 mg subcutaneously at weeks 0, 4 and 16; and placebo at week 12. Patiens assigned to placebo will receive subcutaneous injections of placebo at weeks 0 and 4; then crossover to 45 mg of ustekinumab at weeks 12 and 16. Duration of study participation up to 36 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Must be of Taiwanese or Korean ancestry living in Taiwan or South Korea, respectively
* Have a diagnosis of plaque-type psoriasis at least 6 months prior to first administration of study agent (patients with concurrent psoriatic arthritis may be enrolled)
* Have plaque-type psoriasis covering at least 10% of total body surface area at screening and at the time of first study agent administration
* PASI score of 12 or greater at the time of screening and at time of first study agent administration
* Candidate of phototherapy or systemic treatment of psoriasis (either naïve or history of previous treatment)
* Be able to adhere to the study visit schedule and other protocol requirements
* Capable of giving informed consent prior to any study related procedures.

Exclusion Criteria:

* Currently have a non-plaque form of psoriasis
* Have current drug-induced psoriasis
* Are pregnant or nursing or planning pregnancy (both men and women) while enrolled in the study
* Have used any investigational drug within the previous 4 weeks or 5 times the half life of the investigational agent, whichever is longer
* Have used any biologic within the previous 3 months or 5 times the half life of the biologic, whichever is longer
* Have been hospitalized in the past 3 years for asthma, ever required intubation for treatment of asthma, currently require oral corticosteroids for the treatment of asthma, or required more than one short-term course of oral corticosteroids for asthma within the previous year
* Have a history of latent or active granulomatous infection, including TB, histoplasmosis, or coccidioidomycosis prior to screening.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2008-12; Primary Completion 2009-09 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Centocor, Inc. Clinical Trial, Study Director — Centocor, Inc.
Locations (5):
- South Korea (2):
  - Anyang
  - Seoul
- Taiwan (3):
  - Changhua
  - Kaohsiung County
  - Taipei

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo (CP): Controlled period (Week 0-12) - Placebo Group
- Ustekinumab 45 mg (CP): Controlled period (Week 0-12) - Ustekinumab 45 mg Group
- Placebo -> Ustekinumab 45 mg (After CP): After controlled period (Week 12-36) - receiving Placebo at Weeks 0 and 4 -> receiving ustekinumab 45 mg at Week 12 and Week 16
- Ustekinumab 45 mg (After CP): After controlled period (Week 12-36) - receiving ustekinumab 45 mg at Weeks 0 and 4 -> receiving placebo at Week 12 and ustekinumab 45 mg at Week 16
Period: Controlled Period
Arm/Group | Placebo (CP) | Ustekinumab 45 mg (CP) | Placebo -> Ustekinumab 45 mg (After CP) | Ustekinumab 45 mg (After CP)
Started | 60 | 61 | 0 ("0" in column indicates this reporting group is not relevant to Control Period.) | 0 ("0" in column indicates this reporting group is not relevant to Control Period.)
Completed | 55 | 57 | 0 | 0
Not Completed | 5 | 4 | 0 | 0
Not completed — Adverse Event | 3 | 0 | 0 | 0
Not completed — Lack of Efficacy | 2 | 1 | 0 | 0
Not completed — Other | 0 | 3 | 0 | 0
Period: After Controlled Period
Arm/Group | Placebo (CP) | Ustekinumab 45 mg (CP) | Placebo -> Ustekinumab 45 mg (After CP) | Ustekinumab 45 mg (After CP)
Started | 0 ("0" in column indicates this reporting group is not relevant to after Control Period.) | 0 ("0" in column indicates this reporting group is not relevant to after Control Period.) | 55 | 57 (2 participants discontinued in CP, had follow-up, and are among frequent and serious adverse events.)
Completed | 0 | 0 | 55 | 56
Not Completed | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo (CP) | Ustekinumab 45 mg (CP) | Total
Number analyzed (Participants) | 60 | 61 | 121
Age Continuous [Mean (Standard Deviation); unit: years] | 40.4 (10.06) | 40.9 (12.66) | 40.6 (11.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 11 | 18
  Male | 53 | 50 | 103
Region of Enrollment [Number; unit: participants]
  Republic of Korea | 30 | 31 | 61
  Taiwan | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: The Number of Patients Who Achieved at Least a 75% Improvement in PASI (Psoriasis Area and Severity Index) at Week 12
Description: PASI score can range from 0 (no psoriasis) to 72 (severe psoriasis).
Time Frame: Week 12
Population: Participants were analyzed according to the treatment group to which they were randomized, regardless of the treatment they received.
Measure: Number; unit: Participants
Arm/Group | Placebo | Ustekinumab 45 mg
Number analyzed (Participants) | 60 | 61
Participants | 3 | 41
Statistical Analysis 1: Comparison: Placebo vs Ustekinumab 45 mg; Null Hypothesis: No difference between ustekinumab 45 mg and placebo for the primary endpoint at a significance level of 0.05. With 120 subjects (60 in each treatment group), simulation studies were conducted to calculate the power to detect a treatment difference in the primary endpoint between ustekinumab 45 mg group and placebo using a CMH test stratified by baseline weight (<=65kg vs > 65 kg). For all the scenarios evaluated, the power was > 99% at a significance level of 0.05; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — The study was designed to maintain a Type I error of 0.05 or less for the primary analysis; Stratified by baseline weight (≤ 65 kg vs > 65 kg)

2. Secondary Outcome: The Number of Patients With a Physician's Global Assessment (PGA) Score of Cleared (0) or Minimal (1) at Week 12
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Placebo | Ustekinumab 45 mg
Number analyzed (Participants) | 60 | 61
Participants | 5 | 43
Statistical Analysis 1: Comparison: Placebo vs Ustekinumab 45 mg; Null Hypothesis: No difference between ustekinumab 45 mg and placebo at a significance level of 0.05; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — No multiplicity adjustment was made and nominal p-value was reported; Stratified by baseline weight (≤ 65 kg vs > 65 kg)

3. Secondary Outcome: The Change in Dermatology Life Quality Index (DLQI) From Baseline at Week 12
Description: Scores could range from 0 to 30. A lower DLQI score represents better quality of life.
Time Frame: Baseline to Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | Ustekinumab 45 mg
Number analyzed (Participants) | 60 | 61
Scores on a scale | -0.5 (6.51) | -11.2 (7.07)
Statistical Analysis 1: Comparison: Placebo vs Ustekinumab 45 mg; Null Hypothesis: No difference between ustekinumab 45 mg and placebo at a significance level of 0.05; Test type: Superiority or Other; p < 0.001, ANOVA — No multiplicity adjustment was made and nominal p-value was reported; Analysis of variance on van der Waerden normal scores (Conover, 1980) with treatment and baseline weight (≤ 65kg vs > 65 kg) as factors in the model

ADVERSE EVENTS:
Arm/Group | Placebo (CP) | Ustekinumab 45 mg (CP) | Placebo -> Ustekinumab 45 mg (After CP) | Ustekinumab 45 mg (After CP)
Serious Adverse Events (participants affected / at risk) | 2/60 | 0/61 | 5/55 | 2/59
Other Adverse Events (participants affected / at risk) | 30/60 | 25/61 | 18/55 | 28/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (CP) (N=60) | Ustekinumab 45 mg (CP) (N=61) | Placebo -> Ustekinumab 45 mg (After CP) (N=55) | Ustekinumab 45 mg (After CP) (N=59)
Anal abscess (Infections and infestations) | 1 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 2 | 0
Pulmonary tuberculosis (Infections and infestations) | 0 | 0 | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Muscle injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Henoch-Schonlein purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (CP) (N=60) | Ustekinumab 45 mg (CP) (N=61) | Placebo -> Ustekinumab 45 mg (After CP) (N=55) | Ustekinumab 45 mg (After CP) (N=59)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 3 | 1
Eosinophilia (Blood and lymphatic system disorders) | 2 | 2 | 1 | 3
Injection site erythema (General disorders) | 3 | 0 | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 2 | 0 | 4 | 5
Nasopharyngitis (Infections and infestations) | 3 | 5 | 3 | 8
Upper respiratory tract infection (Infections and infestations) | 7 | 7 | 2 | 5
Hyperglycaemia (Metabolism and nutrition disorders) | 5 | 5 | 3 | 3
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 2 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 16 | 5 | 2 | 4
Psoriasis (Skin and subcutaneous tissue disorders) | 5 | 2 | 3 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less